CLINICAL TRIAL: NCT01989923
Title: Immediate Smoking Cessation for Patients at Risk for Cervical Dysplasia, Cervical Cancer and Lower Genital Tract Dysplasia and Cancer - A Feasibility Study Comparing Nicotine Replacement Therapy With the Electronic Nicotine Delivery System.
Brief Title: Smoking Cessation in Women With Gynecological Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2506
Record Dates: First submitted 2013-07-08; First posted 2013-11-21 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Cervical Dysplasia
Keywords: Smoking cessation; Traditional nicotine replacement therapy; Electronic nicotine delivery devices; electronic cigarettes; cervical dysplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia; Smoking Cessation; Vaping | interventions — Nicotine Replacement Therapy; Transdermal Patch

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nicotine replacement therapy (Active Comparator): Women in this arm of the study will receive 24-hour Nicotine Patches - either 21 mg patches (for 1 pack per day smokers), or 14 mg patches (for 1/2 pack per day smokers) smokers). Patients will use one patch per day for 6 weeks for a total of 42 patches. Women will receive 3 weeks of original strength nicotine patches, and will receive patches half as strong during the last 3 weeks of the study. This will allow for a lower strength of nicotine as each woman continues with smoking cessation.
  Women will also receive nicotine gum or lozenges (subject choice)- these will be 2 mg pieces of nicotine gum or lozenge (approximately 210 pieces). This will account for using 8-10 per day at the beginning of the study and tapering to 2-3 pieces per day by the end of the study.
  Interventions: Other: Nicotine Replacement Therapy
- Electronic Cigarettes (Active Comparator): Women in this arm of the study will receive one "Blu Cig" Electronic Nicotine Delivery Device (E-cigarette) along with 2 electronic cigarette batteries, 1 wall charger and 1 USB charger, cartridges/refills in menthol or regular (patient choice). The number of cartridges is determined by asking each patient the number of packs currently smoked per day, and multiplying 1.5 times the number of packs smoked per day. We plan to decrease the strength of the cartridges by one half after three weeks of intervention. We will give each women supplies and instructions accordingly. This will allow for a lower strength of nicotine as each woman continues with smoking cessation.
  Interventions: Device: Electronic Cigarettes

INTERVENTIONS:
Other: Nicotine Replacement Therapy — Patients will use one patch per day for 6 weeks for a total of 42 patches - they will receive 7 the first visit and then the additional 35 at the second visit. Women will receive 3 weeks of original strength nicotine patches, and will receive patches half as strong during the last 3 weeks of the study. This will allow for a lower strength of nicotine as each woman continues with smoking cessation.
  Other Names: Nicoderm CQ patches (21 or 14 mg patches); Nicorette gum (2 mg); Nicorette lozenges (2 mg)
  Arms: Nicotine replacement therapy
Device: Electronic Cigarettes — The number of cartridges for the electronic cigarettes is determined by asking each patient the number of packs currently smoked per day, and multiplying 1.5 times the number of packs smoked per day. We plan to decrease the strength of the cartridges by one half after three weeks of intervention. We will give each women supplies and instructions accordingly. This will allow for a lower strength of nicotine as each woman continues with smoking cessation
  Other Names: Blu Cig Electronic Nicotine Delivery System
  Arms: Electronic Cigarettes

SUMMARY:
This feasibility study will compare two smoking cessation methods, traditional nicotine replacement therapy and Electronic Nicotine Delivery Systems (electronic cigarettes) in patients with gynecological conditions.

DETAILED DESCRIPTION:
This study will allow women with serious gynecological conditions to sample both traditional nicotine replacement therapy (NRT) and Electronic Nicotine Delivery Systems (electronic cigarettes, ENDS). Whether the woman samples NRT or ENDS first will be randomized. Women will choose the product they wish to try for a 6-week intervention period for smoking cessation. Women choosing NRT will receive a 6-week intervention of a daily nicotine patch plus either nicotine gum or lozenges to use (as needed) throughout the day. The ENDS group will receive an electronic cigarette device with refills to last the 6-week duration of the study. Both groups will receive identical tobacco cessation counseling. As part of the study, each subject will complete a survey conducted at baseline, 6-weeks into the study during intervention, and upon completion of a 6 week follow-up period in which participants receive no intervention. At the 12-week measurement period we will add a qualitative interview that will allow us to ask the women whether the methods were acceptable, caused any problems, and if so, what the problems entailed.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Smokers (defined as those who have smoked at least daily for the last year and who have smoked greater than or equal to 10 or more combustible cigarettes per day during the last year.
* Patients with diagnoses of Cervical Dysplasia, Cervical Cancer and Lower Genital Tract Dysplasia and Cancer
* Ages 18-65 years

Exclusion Criteria:

* Patients unwilling to commit to a 6-week intervention that may include either NRT or ENDS.
* Patients with previous diagnoses of or treatment for cancer - with the exception of non-melanoma skin cancer.
* Presence of any known stroke, heart disease, heart attack, or irregular heart beat.
* Pregnancy and lactation.
* Plan to continue to use other nicotine in addition to the products supplied by the study. These would include: chewing tobacco, snuff, an additional nicotine patch or other nicotine containing products.
* High blood pressure, not well controlled with medication.
* Patients using a non-nicotine "smoking cessation medication."
* Patients taking a prescription medicine for depression or asthma.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2017-04-13 (Actual); Study Completion 2017-04-13 (Actual)

PRIMARY OUTCOMES:
Composite set of questions about the feasibility of successfully using NRT and ENDS over time (assessing change in smoking habits) in Women with Serious Gynecological Conditions | We plan a 3-month study with 6 week follow-up periods.
  To determine the acceptability of traditional nicotine replacement therapy (nicotine patch plus nicotine gum or lozenges) and the ENDS (electronic nicotine delivery system or electronic cigarette as smoking cessation tools in a group of women with cervical dysplasia from the Stephenson Cancer Center Dysplasia Clinics.
  Measurements to assess success:
  1. Reduction of number of cigarettes smoked per day.
  2. Point prevalence abstinence at 7 and 30 days
  3. Smoking cessation rates
  4. Qualitative interviews to assess positives and negatives in these two smoking cessation methods.

SECONDARY OUTCOMES:
Feasibility of Study | 3 months with 6 week follow-up windows
  To determine if we can accure 30 smoking women with cervical dysplasia from the Stephenson Cancer Center for smoking cessation intervention in a 6-month window.

OTHER OUTCOMES:
Product Adherence Diary | Women fill out diary every day for 12 weeks
  The diary will be used for the 6 week intervention portion of the study. This diary is designed to assist individuals in monitoring their smoking and product use during the study. We will encourage each subject to write down every regular cigarette that she smokes as well as every use of the product to which she has been randomized.
Composite set of semi-structured interviews | done at the end of the study (at 12-weeks)
  We will use semi-structured interviews at the 12 week follow-up to help us understand:
  * If the woman currently feels she has a healthy or unhealthy lifestyle, and what factors contribute to this answer.
  * What smoking cessation methods the women have tried in the past, if the methods were acceptable, if they worked, and why or why not.
  * Barriers that might make it difficult for women with this diagnosis to quit smoking using the device they tried in the study.
  * Assists that might make it easier for women with this diagnosis to quit smoking using the device they tried in the study.
  * How the women feel about continuing to use the device that they tried in the trial.
  * Risks the women feel they are taking if they continue to use NRT, ENDS, or decide to return to smoking.
  * What about smoking makes it worth or not worth the risk to these women personally.

CONTACTS AND LOCATIONS:
Overall Officials: Laura A Beebe, PhD, Principal Investigator — University of Oklahoma Health Sciences Center, College of Public Health
Locations (1):
- Stephenson Cancer Center, Oklahoma City, Oklahoma, United States